CLINICAL TRIAL: NCT03109899
Title: Randomized, Controlled Trial of the Sex Pro Mobile App for Young Black MSM in San Francisco and Oakland, CA
Brief Title: Personalized HIV and STI Testing Tool
Acronym: PHASTT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); San Francisco Department of Public Health (Other Government); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Hyman Scott, Medical Director, Clinical Research, Public Health Foundation Enterprises, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-22103; 5K23MH104116 (NIH)
Record Dates: First submitted 2017-03-29; First posted 2017-04-12 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Risk Reduction; HIV; Sexually Transmitted Infections (Not HIV or Hepatitis)
Keywords: mHealth; HIV Prevention
MeSH Terms: conditions — Risk Reduction Behavior; Sexually Transmitted Diseases; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this arm will have access to the Sex Pro mobile app and support for HIV/STI testing and PrEP uptake.
  Interventions: Behavioral: Sex Pro mobile Application
- Control (No Intervention): Participants in this arm will be given the local standard of care for HIV/STI testing and PrEP access.

INTERVENTIONS:
Behavioral: Sex Pro mobile Application — Mobile mHealth app that provides HIV risk assessment, home HIV/STI testing options, and PrEP uptake support for young Black MSM.
  Arms: Intervention

SUMMARY:
The PHASTT Study is focused on understanding of facilitators and barriers to mHealth use among young Black men who have sex with men (MSM), and testing a novel mobile app to increase HIV/STI testing and PrEP uptake.

DETAILED DESCRIPTION:
The Sex Pro mobile application (app) being tested facilitates home HIV-testing, home sexually transmitted infection (STI) test self-collection, and pre-exposure prophylaxis (PrEP) uptake. The app integrates a personalized HIV risk assessment with home HIV and STI testing options for young, Black MSM.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black.
* Self-report being HIV negative.
* Report anal sex with at two or more male sex partners in the prior 12 months.
* Own an iOS or Android mobile phone.
* Willing and able to give written informed consent to participate in all activities outlined by the protocol.

Exclusion Criteria:

* Inadequate contact information for follow-up
* In a mutually monogamous sexual relationship for the past 12 months
* Currently taking PrEP
* Does not have reliable access to the internet
* Does not live, work or play in the San Francisco Bay Area
* Currently enrolled in another HIV intervention study
* Prior enrollment in an HIV vaccine trial with receipt of experimental vaccine product
* Any medical, psychiatric, or social condition, or occupational, or other responsibility that, in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 80 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
The feasibility and acceptability of Sex Pro to increase HIV/STI testing and PrEP uptake among young Black MSM. | 9 months
  As measured via computer assisted interview (CASI)

SECONDARY OUTCOMES:
The rate of HIV testing in the Sex Pro mobile application intervention versus control arms. | 9 months
  As measured by CASI
The rate of STI testing in the Sex Pro mobile application intervention versus control arms. | 9 months
  As measured by CASI
The rate of PrEP uptake in the Sex Pro mobile application intervention versus control arms. | 9 months
  As measured by pharmacy confirmation
Changes in sexual risk behaviors among young Black MSM in the Sex Pro mobile application intervention vs. control arms | 9 months
  As measured via CASI

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Scott, Principal Investigator — Public Health Foundation Enterprises; San Francisco Department of Public Health
Locations (1):
- Bridge HIV, San Francisco Department of Public Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No